CLINICAL TRIAL: NCT02180711
Title: An Open-label, Phase 1b/2 Study of Acalabrutinib Alone or in Combination Therapy in Subjects With B-cell Non-Hodgkin Lymphoma
Brief Title: Study of Acalabrutinib Alone or in Combination Therapy in Subjects With B-cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-003; 2023-509350-63-00 (Registry Identifier: CTIS (EU)); 2019-000111-84 (EudraCT Number)
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Bruton tyrosine kinase inhibitor; Btk; Follicular Lymphoma; FL; acalabrutinib; ACP-196; MZL; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — acalabrutinib; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: acalabrutinib Regimen 1 (Experimental): acalabrutinib Regimen 1 for relapsed, refractory Follicular Lymphoma subjects
  Interventions: Drug: acalabrutinib
- Part 1: acalabrutinib Regimen 2 (Experimental): acalabrutinib Regimen 2 + rituximab for relapsed, refractory, or treatment naive Follicular Lymphoma subjects
  Interventions: Drug: acalabrutinib; Drug: rituximab (IV)
- Part 2: acalabrutinib Regimen 1 (Experimental): acalabrutinib Regimen 1 for relapsed, refractory Marginal Zone Lymphoma subjects
  Interventions: Drug: acalabrutinib
- Part 2: acalabrutinib Regimen 2 (Experimental): acalabrutinib Regimen 2 + rituximab for relapsed, refractory Marginal Zone Lymphoma subjects
  Interventions: Drug: acalabrutinib; Drug: rituximab (IV)
- Part 3: acalabrutinib Regimen 1 (Experimental): acalabrutinib Regimen + lenalidomide + rituximab for relapsed, refractory Follicular Lymphoma subjects
  Interventions: Drug: acalabrutinib; Drug: rituximab (IV); Drug: Lenalidomide

INTERVENTIONS:
Drug: acalabrutinib
  Other Names: ACP-196
Drug: rituximab (IV)
  Arms: Part 1: acalabrutinib Regimen 2; Part 2: acalabrutinib Regimen 2; Part 3: acalabrutinib Regimen 1
Drug: Lenalidomide
  Arms: Part 3: acalabrutinib Regimen 1

SUMMARY:
Part 1: To characterize the safety profile of acalabrutinib alone or in combination with rituximab in subjects with R/R FL.

Part 2: To characterize the activity of acalabrutinib alone or in combination with rituximab in subjects with R/R MZL, as measured by ORR.

Part 3: To characterize the safety of acalabrutinib in combination with rituximab and lenalidomide in subjects with R/R FL

DETAILED DESCRIPTION:
An Open-label, Phase 1b/2 Study of Acalabrutinib Alone or in Combination Therapy in Subjects with B-cell Non-Hodgkin Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Part 1: A confirmed diagnosis of FL Grade 1, 2, or 3a, which has relapsed after, or been refractory to ≥ 1 prior therapy for FL, or subjects who have not previously received systemic anticancer therapy for FL., and which requires treatment.
* Part 2: For subject with relapsed or refractory MZL:

Histologically confirmed MZL including splenic, nodal, and extranodal sub-types

1. Subjects with splenic MZL must have an additional measurable lesion, nodal or extranodal, as described in inclusion criterion #4;
2. Subjects with gastric mucosa-associated lymphoid tissue (MALT) lymphoma must be Helicobacter pylori (HP)-negative

   * Part 3: For subjects with FL: Pathologically confirmed diagnosis of FL Grade 1, 2, or 3a, which has relapsed after, or been refractory to ≥ 1 prior therapy for FL and which requires treatment per National Cancer Institute or ESMO clinical practice guidelines.
   * Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
   * Agreement to use contraception during the study and for 30 days after the last dose of study drugs if sexually active and able to bear or beget children.

Exclusion Criteria:

* •A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or Qtc >480 msec
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, gastric bypass, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Breast feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2028-12-29 (Estimated)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (24):
  - Research Site, Tucson, Arizona
  - Research Site, Downey, California
  - Research Site, Duarte, California
  - Research Site, Fountain Valley, California
  - Research Site, Santa Monica, California
  - Research Site, Coral Gables FL, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Ann Arbor, Michigan
  - Research Site, Morristown, New Jersey
  - Research Site, Hawthorne, New York
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, Columbus, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Spokane, Washington
  - Research Site, Waukesha, Wisconsin
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
- Italy (3):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Palermo

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-003&attachmentIdentifier=9c32d093-ff79-4c9c-8964-d247ffdc898d&fileName=ace-ly-003-csp-v8_CCI_redacted_Redacted_pdfa.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-003&attachmentIdentifier=e5e76973-610b-4e50-a5bd-c08b2dcdac03&fileName=ace-ly-003-sap-ed-1-part-2-3_redacted_Redacted_pdfa.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-003&attachmentIdentifier=dd36939a-2abe-4257-980d-f7824334df84&fileName=ace-ly-003-study-synopsis-part-2-3_CCI_redacted_Redacted_pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- P1: RR Acalabrutinib 100 mg BID: (Relapsed/Refractory Cohort: Acalabrutinib 100 mg Twice a Day (BID))
- P1: RR Acalabrutinib 100 mg BID + Rituximab: (Relapsed/Refractory Cohort: Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2)
- P1: RR Acalabrutinib 200 mg QD: (Relapsed/Refractory Cohort: Acalabrutinib 200 mg once a day (QD))
- P1: TN Acalabrutinib 100 mg BID + Rituximab: (Treatment Naive Cohort: Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2)
- P2: Acalabrutinib: (Acalabrutinib 100 mg Twice a Day (BID))
- P2: Acalabrutinib + Rituximab: (Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2)
- P3: Acalabrutinib + Rituximab + Lenalidomide 15 mg: (Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2 + Lenalidomide 15 mg Daily (QD))
- P3: Acalabrutinib + Rituximab + Lenalidomide 20 mg: (Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2 + Lenalidomide 20 mg Daily (QD))
Period: Overall Study
Arm/Group | P1: RR Acalabrutinib 100 mg BID | P1: RR Acalabrutinib 100 mg BID + Rituximab | P1: RR Acalabrutinib 200 mg QD | P1: TN Acalabrutinib 100 mg BID + Rituximab | P2: Acalabrutinib | P2: Acalabrutinib + Rituximab | P3: Acalabrutinib + Rituximab + Lenalidomide 15 mg | P3: Acalabrutinib + Rituximab + Lenalidomide 20 mg
Started | 12 | 13 | 2 | 13 | 43 | 1 | 8 | 21
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 13 | 2 | 13 | 43 | 1 | 8 | 21
Not completed — Death | 0 | 1 | 0 | 0 | 7 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 4 | 3 | 0 | 3 | 2
Not completed — - Disease Progression | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — - Subject Started Alternative Cancer Therapy | 7 | 6 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — - Study Terminated by Sponsor | 2 | 3 | 0 | 5 | 32 | 0 | 4 | 13
Not completed — - Enrolled into Follow-up Study | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — - Other | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The All-treated Population, defined as all subjects who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | P1: RR Acalabrutinib 100 mg BID | P1: RR Acalabrutinib 100 mg BID + Rituximab | P1: RR Acalabrutinib 200 mg QD | P1: TN Acalabrutinib 100 mg BID + Rituximab | P2: Acalabrutinib | P2: Acalabrutinib + Rituximab | P3: Acalabrutinib + Rituximab + Lenalidomide 15 mg | P3: Acalabrutinib + Rituximab + Lenalidomide 20 mg | Total
Number analyzed (Participants) | 12 | 13 | 2 | 13 | 43 | 1 | 8 | 21 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (16.0) | 66.7 (10.6) | 59.0 (21.2) | 59.6 (12.2) | 66.0 (10.0) | 43.0 (NA) — There was only one participant in this treatment group. | 62.5 (9.7) | 63.0 (9.7) | 64.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 1 | 8 | 17 | 1 | 1 | 6 | 48
  Male | 6 | 5 | 1 | 5 | 26 | 0 | 7 | 15 | 65
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 1 | 1 | 0 | 3 | 3 | 10
  Not Hispanic or Latino | 12 | 11 | 2 | 12 | 41 | 1 | 5 | 17 | 101
  Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Black or African American | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 7
  Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  White | 11 | 13 | 2 | 12 | 38 | 1 | 7 | 17 | 101
Region of Enrollment [Number; unit: Participants]
  Canada | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 9
  Italy | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
  United States | 12 | 13 | 2 | 13 | 36 | 1 | 8 | 16 | 101

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Incidence of Treatment-emergent Adverse Events.
Description: Treatment-emergent adverse events were used to characterize the safety profile of acalabrutinib alone or in combination with rituximab in participants with relapsed/refractory follicular lymphoma (R/R FL).
Time Frame: From the first dose of study drug until study discontinuation, 30 days after the last dose of study drug or one day before the first subsequent anticancer therapy, whichever was earlier, up to 80.7 months (the maximum participant's time on this study).
Measure: Number; unit: Number of participants
Groups:
- Part 1: Acalabrutinib 100 mg BID: (Relapsed/Refractory Cohort: Acalabrutinib 100 mg Twice a Day (BID))
- Part 1: Acalabrutinib 100 mg BID + Rituximab: (Relapsed/Refractory Cohort: Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2)
- Part 1: Relapsed or Refractory Acalabrutinib 200 mg QD: (Relapsed/Refractory Cohort: Acalabrutinib 200 mg once a day (QD))
- Part 1: Acalabrutinib 100 mg Rituximab: (Treatment Naive Cohort: Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2)
Arm/Group | Part 1: Acalabrutinib 100 mg BID | Part 1: Acalabrutinib 100 mg BID + Rituximab | Part 1: Relapsed or Refractory Acalabrutinib 200 mg QD | Part 1: Acalabrutinib 100 mg Rituximab
Number analyzed (Participants) | 12 | 13 | 2 | 13
Number of participants | 12 | 13 | 2 | 13

2. Primary Outcome: Part 2: Investigator Assessed Objective Response Rate (ORR) According to the Lugano Classification for Non-Hodgkin Lymphoma (NHL).
Description: The objective response rate (ORR) is used to characterize the activity of acalabrutinib alone or in combination with rituximab in participants with relapsed/refractory marginal zone lymphoma (R/R MZL).
Time Frame: Based on all response assessments since the first dose of study drug until study discontinuation or the initiation of subsequent anticancer therapy, whichever was earlier, up to 65.1 months (the maximum participant's time on this study).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part 2: Acalabrutinib: (Acalabrutinib 100 mg Twice a Day (BID))
- Part 2: Acalabrutinib + Rituximab: (Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2)
Arm/Group | Part 2: Acalabrutinib | Part 2: Acalabrutinib + Rituximab
Number analyzed (Participants) | 43 | 1
Percentage of participants | 60.5 [44.4 to 75.0] | 0 [0 to 97.5]

3. Primary Outcome: Part 3: Incidence of Treatment-emergent Adverse Events.
Description: Treatment-emergent adverse events were used to characterize the safety of acalabrutinib in combination with rituximab and lenalidomide in participants with relapsed/refractory follicular lymphoma (R/R FL).
Time Frame: From the first dose of study drug until study discontinuation, 30 days after the last dose of study drug or one day before the first subsequent anticancer therapy, whichever was earlier, up to 54.3 months (the maximum participant's time on this study).
Measure: Number; unit: Number of participants
Groups:
- Part 3: Acalabrutinib + Rituximab + Lenalidomide 15 mg: (Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2 + Lenalidomide 15 mg Daily (QD))
- Part3: Acalabrutinib + Rituximab + Lenalidomide+20mg: (Acalabrutinib 100 mg Twice a Day (BID) + Rituximab 375 mg/m2 + Lenalidomide 20 mg Daily (QD))
Arm/Group | Part 3: Acalabrutinib + Rituximab + Lenalidomide 15 mg | Part3: Acalabrutinib + Rituximab + Lenalidomide+20mg
Number analyzed (Participants) | 8 | 21
Number of participants | 8 | 21

ADVERSE EVENTS:
Time Frame: Treatment-emergent period, i.e. from the first dose of study drug until study discontinuation, 30 days after the last dose of study drug, or one day before the initiation of the subsequent anticancer therapy, whichever occurred earlier, up to 80.7 months for part 1, up to 65.1 months for part 2, and up to 54.3 months for part 3.
Description: Adverse events are coded per MedDRA version 25.0 for Part 1. Adverse events are coded per MedDRA version 26.1 for Part 2 and Part 3.
Arm/Group | P1: RR Acalabrutinib 100 mg BID | P1: RR Acalabrutinib 100 mg BID + Rituximab | P1: RR Acalabrutinib 200 mg QD | P1: TN Acalabrutinib 100 mg BID + Rituximab | P2: Acalabrutinib | P2: Acalabrutinib + Rituximab | P3: Acalabrutinib + Rituximab + Lenalidomide 15 mg | P3: Acalabrutinib + Rituximab + Lenalidomide 20 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/13 | 0/2 | 0/13 | 7/43 | 0/1 | 1/8 | 3/21
Serious Adverse Events (participants affected / at risk) | 2/12 | 5/13 | 0/2 | 3/13 | 9/43 | 1/1 | 4/8 | 11/21
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13 | 2/2 | 13/13 | 41/43 | 1/1 | 8/8 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1: RR Acalabrutinib 100 mg BID (N=12) | P1: RR Acalabrutinib 100 mg BID + Rituximab (N=13) | P1: RR Acalabrutinib 200 mg QD (N=2) | P1: TN Acalabrutinib 100 mg BID + Rituximab (N=13) | P2: Acalabrutinib (N=43) | P2: Acalabrutinib + Rituximab (N=1) | P3: Acalabrutinib + Rituximab + Lenalidomide 15 mg (N=8) | P3: Acalabrutinib + Rituximab + Lenalidomide 20 mg (N=21)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 2 (3)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1: RR Acalabrutinib 100 mg BID (N=12) | P1: RR Acalabrutinib 100 mg BID + Rituximab (N=13) | P1: RR Acalabrutinib 200 mg QD (N=2) | P1: TN Acalabrutinib 100 mg BID + Rituximab (N=13) | P2: Acalabrutinib (N=43) | P2: Acalabrutinib + Rituximab (N=1) | P3: Acalabrutinib + Rituximab + Lenalidomide 15 mg (N=8) | P3: Acalabrutinib + Rituximab + Lenalidomide 20 mg (N=21)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 5 (15) | 4 (6) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (6) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 4 (6) | 1 (2) | 5 (6) | 5 (5) | 0 (0) | 1 (1) | 6 (7)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 8 (8)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 5 (9) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (15) | 1 (1) | 1 (1) | 2 (3)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (16) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (11) | 0 (0) | 1 (3) | 7 (11)
Platelet count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 3 (5)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (6) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (3) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 0 (0) | 5 (7) | 6 (6) | 0 (0) | 1 (1) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4) | 0 (0) | 3 (3) | 6 (7) | 0 (0) | 3 (3) | 3 (3)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc annular tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 1 (1) | 2 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 7 (11) | 0 (0) | 2 (7) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudoxanthoma elasticum (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (14) | 5 (8) | 0 (0) | 6 (8) | 15 (18) | 1 (1) | 3 (4) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 7 (14) | 0 (0) | 2 (2) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 3 (3) | 0 (0) | 1 (2) | 10 (13) | 0 (0) | 3 (3) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 5 (6) | 1 (1) | 1 (1) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Tympanosclerosis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 3 (3) | 1 (1) | 3 (3) | 6 (8)
Hyperprolactinaemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (8) | 0 (0) | 2 (2) | 5 (11)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (5) | 5 (7) | 0 (0) | 1 (3) | 4 (8)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypogonadism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (12) | 0 (0) | 2 (4) | 5 (12) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (3) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Eyelid bleeding (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleral hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 4 (5) | 0 (0) | 0 (0) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0) | 3 (8) | 7 (8) | 0 (0) | 1 (1) | 5 (6)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (11) | 5 (11) | 1 (1) | 7 (19) | 12 (14) | 1 (4) | 4 (6) | 12 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (4) | 3 (4) | 0 (0) | 1 (1) | 9 (24)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 5 (8) | 1 (1) | 4 (8) | 15 (18) | 0 (0) | 0 (0) | 8 (12)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 4 (6) | 0 (0) | 1 (1) | 2 (10)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 4 (4) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 5 (7)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (11) | 8 (12) | 0 (0) | 7 (15) | 15 (25) | 0 (0) | 3 (3) | 7 (13)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 4 (8) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 5 (6)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (6) | 0 (0) | 2 (2) | 3 (3) | 1 (4) | 2 (2) | 5 (5)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 6 (8)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02180711/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT02180711/SAP_001.pdf